CLINICAL TRIAL: NCT07398508
Title: Phase I/II Study of NORTHERA (DROXIDOPA) for Dysautonomia in Pediatric Survivors of Menkes Disease: Double-blind Placebo-controlled Randomized Crossover Clinical Trial.
Brief Title: Phase I/II Study of NORTHERA (DROXIDOPA) for Dysautonomia in Pediatric Survivors of Menkes Disease.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stephen G. Kaler (Other)
Responsible Party: Sponsor-Investigator, Stephen G. Kaler, Professor, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ACYY0326
Record Dates: First submitted 2026-02-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Menkes Disease
Keywords: Menkes disease, dysautonomia, orthostatic hypotension
MeSH Terms: conditions — Menkes Kinky Hair Syndrome; Autonomic Nervous System Diseases; Hypotension, Orthostatic | interventions — Droxidopa

STUDY DESIGN:
Intervention Model Description: Double-blind Placebo-controlled Randomized Crossover Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Droxidopa Treatment Arm (Experimental): Oral administration of droxidopa study drug.
  Interventions: Drug: Droxidopa Oral Product
- Placebo Control Arm (Placebo Comparator): Oral administration of placebo control capsules that are indistinguishable from study drug.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: Droxidopa Oral Product — 1 month supply will contain pre-prepared capsules containing either 20mg, 40mg, or 60mg Droxidopa, plus 300 ml of simple syrup. For each dose, add the contents of 1 capsule and 10 ml of simple syrup to a plastic 1 ounce medication cup. Simple syrup will be dispensed from a larger bottle using a 10mL syringe. Mix by swirling briefly and consume the entire contents. Prepare the suspension freshly for each dose and take the prescribed dose twice daily, at approximately 8am and 2pm.
  Other Names: NORTHERA
  Arms: Droxidopa Treatment Arm
Other: Placebo Control — 1 month supply will contain pre-prepared capsules containing cellulose microcrystalline placebo, plus 300 ml of simple syrup. For each dose, add the contents of 1 capsule and 10 ml of simple syrup to a plastic 1 ounce medication cup. Simple syrup will be dispensed from a larger bottle using a 10mL syringe. Mix by swirling briefly and consume the entire contents. Prepare the suspension freshly for each dose and take the prescribed dose twice daily, at approximately 8am and 2pm.
  Other Names: Placebo pill
  Arms: Placebo Control Arm

SUMMARY:
This clinical trial will evaluate the safety, tolerability, dosing, and efficacy of Northera (Droxidopa) in children with Menkes disease aged 7 to 17 years who survived the major neurodegenerative and neurocognitive effects of Menkes disease through early Copper Histidinate treatment. The investigator hypothesizes that Northera (Droxidopa) treatment in pediatric Menkes disease survivors with symptoms of dysautonomia (e.g., syncope, dizziness, orthostatic hypotension, abnormal sinoatrial conduction, and bowel or bladder dysfunction) from deficiency of the cuproenzyme, dopamine-beta-hydroxylase, will be safe and will correct or improve blood neurochemical levels, raise systolic blood pressure, and produce symptomatic improvement and a better quality of life. The investigator will test this hypothesis, in six to ten child or adolescent Menkes disease survivors through a placebo-controlled trial to evaluate adverse event rates and whether oral administration of Northera (Droxidopa) at doses established for individual subjects by careful dose titration improves plasma norepinephrine and dihydroxyphenylglycol (DHPG) levels, raises systolic blood pressure, and improves performance on tests of physical exertion. As an exploratory outcome measure, the study will validate the Orthostatic Hypotension Symptom Assessment (OHSA) questionnaire for this population for two four-week periods of either active or placebo treatment.

Aim 1. Determine the safety of Droxidopa in Menkes disease pediatric survivors.

Aim 2. Determine the efficacy of Droxidopa in Menkes disease survivors. The investigator hypothesizes that low-dose Droxidopa treatment in classic Menkes disease survivors aged 7 to 17 will improve orthostatic hypotension and ameliorate other signs and symptoms of dysautonomia. This pilot study will employ an ascending dose paradigm in a double-blind placebo-controlled randomized crossover design to optimize statistical power and rigorously discern treatment effects on 1) tilt table tests of orthostatic hypotension, 2) systolic and diastolic blood pressure, 3) plasma neurochemical levels and 4) tests of physical exertion. The trial will also validate the Orthostatic Hypotension Symptom Assessment (OHSA) questionnaire for this population of children and adolescents. This study addresses an important unmet clinical need for subjects with a rare disease, Menkes disease.

DETAILED DESCRIPTION:
This proposal outlines a concerted effort to evaluate the safety and efficacy of the synthetic amino acid L-threo-3,4-dihydroxyphenylserine (Droxidopa) for the symptoms of dysautonomia that are common in pediatric survivors of Menkes disease. Classic Menkes disease is a fatal X-linked recessive disorder of copper homeostasis that results from variants in a copper transporter gene, ATP7A, and has an estimated birth prevalence of 1 in 35,000 males. The tragedy of Menkes disease involves the apparent good health of affected infants both prenatally and during the first 6-8 weeks of life, after which signs and symptoms of central nervous system (CNS) degeneration emerge. Our prior clinical research demonstrated that early diagnosis (within approximately 28 days of birth) and three years of daily treatment with subcutaneous injections of Copper Histidinate (NDA #34,166) can extend survival and markedly improve neurodevelopmental and neurocognitive outcomes. However, survivors of the illness's severe CNS effects often develop symptoms of dysautonomia, such as syncope, dizziness, orthostatic hypotension, abnormal sinoatrial conduction, nocturnal bradycardia, and bowel or bladder dysfunction beginning in middle childhood. These problems are caused by partial deficiency of dopamine-beta-hydroxylase (DBH), which requires ATP7A to deliver Cu to intracellular compartments for incorporation as its enzymatic cofactor. DBH normally converts dopamine to norepinephrine, and similar symptoms are reported in individuals with congenital absence of DBH, an autosomal recessive disorder. The drug Droxidopa is a synthetic amino acid L-threo-3,4-dihydroxyphenylserine and can be metabolized by the non-copper dependent enzyme DOPA decarboxylase to produce norepinephrine, bypassing the DBH enzymatic defect. The investigator has demonstrated neurochemical improvements in a mouse model of Menkes disease with this compound, as well as in adult Menkes disease survivors over age 18 in a detailed trial (NCT04977388). The investigator recently developed a new liquid suspension of Droxidopa to test smaller doses in pediatric survivors of Menkes disease in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Children or adolescents with Menkes disease who survived beyond the expected natural history, attained independent ambulation, and attend school after early CuHis treatment for three years, who manifest clinical signs and symptoms of dysautonomia, e.g., orthostatic hypotension: specifically, a decrease in systolic or diastolic blood pressure of at least 20 or 10 mm Hg, respectively, within three minutes after standing, and/or chronic diarrhea: production of loose stools with or without increased stool frequency for more than four weeks immediately preceding enrollment.
2. History of at least thrice weekly occurrence of dizziness/feeling lightheaded while standing upright and/or thrice weekly episodes of diarrhea or an urgent need to defecate after food ingestion for more than four weeks immediately preceding enrollment.
3. Documented mutation in ATP7A.
4. One parent must sign and date an Informed Consent Form (ICF) and patient must also assent.
5. Age 7 to 17 years. (Enrollment will be staggered so that at least the first two children enrolled are aged 12-17 years.)
6. Ability to adhere to the prescribed oral Northera (Droxidopa) regimen.
7. Willingness to comply with all study visits and procedures.

Exclusion Criteria:

1. Pre-existing liver (e.g., hepatitis, biliary atresia, cirrhosis) or kidney disease (i.e., calculated glomerular filtration rate <30 ml/min).
2. History of age-adjusted stage 1 hypertension (≥ 95th percentile) [1] (Also see Attachment A).
3. History of anti-hypertensive therapy, heart failure (or decreased ejection fraction), cardiac arrhythmia, or bleeding diatheses.
4. Any disease or condition that, in the opinion of the Investigator, has a high probability of precluding the subject from completing the study or where the subject cannot or will not appropriately comply with study requirements.
5. Any alpha-1 adrenoreceptor agonist, beta-blocker, DOPA decarboxylase inhibitor, midodrine, ephedrine, or any triptan medication as a concomitant medication.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of SAEs | 10 weeks
  This is to measure safety and tolerability of study drug in children and adolescents with Menkes disease. The study will determine the adverse event profile of the formulation by comparing the time-to-event of serious adverse events (SAEs) and adverse events (AEs) between treatment and placebo arms as defined in the protocol.

SECONDARY OUTCOMES:
Change in level of plasma norepinephrine and dihydroxyphenylglycol after Northera (Droxidopa) | Baseline and post intervention at 4 weeks
  Plasma L-DOPS levels: Levels of L-threo-3,4-dihydroxyphenylserine (L-DOPS, droxidopa) may be measured for comparison to the known pharmacokinetic (PK) profile of Northera (Droxidopa) (peak level at approximately 3 hrs). The assay for plasma LDOPS and plasma catecholamines (High Performance Liquid Chromatography with electrochemical detection) is the same. Measurements of L-DOPS may permit correlation between plasma L-DOPS and plasma norepinephrine levels.
Change in systolic blood pressure | Baseline and post intervention at 4 weeks
  Blood pressure (BP) will be measured using a standard blood pressure monitor while subjects are standing, and between supine and head-up tilt table positions after Northera (Droxidopa). Unit: mm Hg. Tilt Table testing involves positioning a patient onto the tilt table with feet resting on footplates. Continuous blood pressure monitors are then attached to the subject. The entire table can be tilted to move from 0˚ to 60˚angle in approximately 45s, allowing determination of changes in pulse and blood pressure based on supine (0˚) and standing (60˚) positions.
Average number of daily bowel movements | Baseline, 4 weeks
  Gastrointestinal symptoms will be monitored using irritable bowel syndrome-diarrhea report. Decreased daily bowel movements counts as an improvement.
Average time standing | Baseline and post intervention at 4 weeks
  This is to measure any improvement in physicality using performance of physical exertion tests. The longer the time standing, the greater the improvement. Unit: minutes.
Average 6-minute walk distance | Baseline and post intervention at 4 weeks
  This is to measure any improvement in physicality using performance of physical exertion tests. The further the distance, the greater the improvement. The primary measurement taken from a 6-minute walk test (6MWT) is the final distance someone manages to walk, which we refer to as the 6MWD (6-minute walk distance), which can be used to assess a patient's functional status. For everyday healthy people, the average distance walked during this test is between 400 and 700 meters.

OTHER OUTCOMES:
Change in scores on the Orthostatic Hypotension Symptom Assessment questionnaire after Northera (Droxidopa) | Baseline and post intervention at 4 weeks
  The Orthostatic Hypotension Questionnaire (OHQ) was developed, with two components: the six-item symptoms assessment scale and a four-item daily activity scale to assess the burden of symptoms. Validation analyses were then performed on the two scales and a composite score of the OHQ. Lower the OHQ scores, less severe the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Kaler, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Vagelos College of Physicians and Surgeons, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided